CLINICAL TRIAL: NCT02569307
Title: A Randomised Double Blind Placebo Controlled Pilot Study of Minocycline and/or Omega-3 Fatty Acids Added to Treatment as Usual for At Risk Mental States
Brief Title: Minocycline and/or Omega-3 Fatty Acids Added to Treatment as Usual for At Risk Mental States
Acronym: NAYAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PILL-NAYAB-001
Record Dates: First submitted 2015-10-03; First posted 2015-10-06 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: At Risk Mental State (ARMS); Psychosis
Keywords: At Risk of Mental State; Prodromal Phase; Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Minocycline; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Minocycline (Active Comparator): Minocycline added to TAU Minocycline will be administered in 200mg once daily dose
  Interventions: Drug: Minocycline
- Omega-3 fatty acids (Active Comparator): Omega-3 fatty acids added to TAU Omega-3 fatty acids will be administered in 1.2mg once daily dose
  Interventions: Drug: Omega-3 fatty acids
- Placebo (Active Comparator): Placebo added to TAU
  Interventions: Drug: Placebo
- Minocycline Plus Omega-3 fatty acids (Active Comparator): Minocycline+Omega-3 fatty acids added to TAU ,Minocyline will be administered in 200mg once daily dose and Omega-3 fatty acids 1.2 g taken as once daily dose
  Interventions: Drug: Minocycline Plus Omega-3 fatty acids

INTERVENTIONS:
Drug: Minocycline — Minocycline added to TAU Minocycline will be administered in 200mg once daily dose
  Arms: Minocycline
Drug: Omega-3 fatty acids — Omega-3 fatty acids added to TAU Omega-3 fatty acids will be administered in 1.2g once daily dose
  Arms: Omega-3 fatty acids
Drug: Placebo — Placebo added to TAU
  Arms: Placebo
Drug: Minocycline Plus Omega-3 fatty acids — Minocycline will be administered in 200mg once daily dose and Omega-3 fatty acid 1.2g taken as once daily dose
  Arms: Minocycline Plus Omega-3 fatty acids

SUMMARY:
This is a randomized double-blind placebo controlled trial which aims to evaluate the efficacy and tolerability of minocycline and Omega-3 fatty acids for patients with ARMS. Specifically to determine whether the addition of minocycline and / or Omega-3 fatty acids to Treatment as Usual in an operationalized ARMS population in Pakistan:

DETAILED DESCRIPTION:
Primary hypothesis is that the persons with ARMS who are prescribed minocycline and / or Omega-3 fatty acids will have reduced transition rates to psychosis over a one year follow up period (from baseline) compared with Treatment-As-Usual (TAU). The transition rates will be lowest in the group receiving minocycline and Omega-3 fatty acids in combination.

Secondary objective is to determine that the Persons with ARMS who are prescribed minocycline and / or Omega-3fatty acids in combination will have greatest symptom reduction compared with TAU.

This study will be a six-month intervention of minocycline and/or Omega-3 fatty acids added to TAU in patients with ARMS, using a randomised, placebo-controlled, double-blind factorial design.The study will be a four-arm trial: one arm will receive minocycline with TAU; the second arm will receive Omega-3 fatty acids with TAU; the third arm will receive both minocycline and Omega-3 fatty acids with TAU; the fourth arm will receive placebo with TAU.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female help seeking individuals aged between 16-35 years.
2. Meets at least one of the criteria for ARMS (see CAARMS Operationalized Intake Criteria section below).
3. Assessed as competent to provide informed consent.

Exclusion Criteria:

1. History ofpreviously experiencing a psychotic illness (treated or untreated).
2. IQ < 70 and/or history of learning disability.
3. Any pre-existing inflammatory conditions e.g. rheumatoid arthritis.
4. Organic brain disease e.g. epilepsy.
5. treatment with an antipsychotic or mood-stabilising agent.
6. Prior history of intolerance or serious side effects (hepatotoxicity, photosensitivity, blood dyscrasias) to any of the tetracyclines or Omega-3 fatty acids.
7. Concomitant penicillin therapy or concomitant anticoagulant therapy.
8. Active substance abuse (except nicotine or caffeine) or dependence within the last three months, according to DSM-V criteria.
9. Treatment with warfarin or lamotrigine.
10. Current or previous treatment with tetracycline antibiotics or Omega-3 fatty acids in the preceding three months before study entry.
11. Current treatment with any anti-inflammatory medication.
12. Treatment with electroconvulsive therapy within the 12 weeks preceding the study.
13. Active expression of suicidal ideation (CAARMS item 7.3 severity score 6) or current aggression/dangerous behaviour (CAARMS item 5.4 severity score 6). 14. Relevant current or past hematologic, hepatic, renal, neurological or other medical disorder that in the opinion of the principal investigator may interfere with the study.

15. Pregnant or breastfeeding females.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 326 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Transition to psychotic disorder | 12 Months
  Structure Clinical interview for DSM-IV(SCID) (Michael B et al,. 2002) to confirm the transition to psychosis.

SECONDARY OUTCOMES:
Measured severity ofAt Risk of Mental State ( ARMS) symptoms | 12 Months
  Comprehensive Assessment of At-Risk Mental States (CAARMS) (Berger, GEet al2006).A semi-structured interview that assists in the identification of individuals at risk of developing a first-episode psychotic disorder and measured the severity of ARMS symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Inti Qurashi, MD, Principal Investigator — Manchester University ,UK
Locations (7):
- Pakistan (7):
  - Abasi Shaheed Hospital, Karachi, Sindh
  - Civil hospital Karachi, Karachi, Sindh
  - Karwn e Hayat, Karachi, Sindh
  - Colleges and Universities, Karachi, Sindh
  - Community, Karachi, Sindh
  - General Practitioners (GPs), Karachi, Sindh
  - Institute of Behavioral Sciences, Karachi, Sindh

REFERENCES:
- [Derived] Qurashi I, Chaudhry IB, Khoso AB, Farooque S, Lane S, Husain MO, Chu S, Sarginson J, Hamarani M, Naqvi HA, Razzaque B, Minhas FA, Yung AR, Deakin JFW, Husain N. A randomised, double-blind, placebo-controlled trial of minocycline and/or omega-3 fatty acids added to treatment as usual for at-risk mental states (NAYAB): study protocol. Trials. 2017 Nov 9;18(1):524. doi: 10.1186/s13063-017-2275-y. PMID 29121974
- See also: Website of Pakistan Institute of Learning and Living — http://pill.org.pk